CLINICAL TRIAL: NCT01593475
Title: A Phase II Study of Induction Chemotherapy With Gemcitabine and Cisplatin Followed by Concurrent Chemoradiotherapy for Locally Advanced Unresectable Pancreatic Carcinoma
Brief Title: Induction Chemotherapy With Gemcitabine and Cisplatin Followed by CCRT for Unresectable Pancreatic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Woojin Lee, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-567
Record Dates: First submitted 2012-05-01; First posted 2012-05-08 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Carcinoma Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction chemotherapy followed by CCRT (Experimental): In one cycle (4-weeks), gemcitabine 1,000 mg/m2 will be given by 30-minute intravenous infusion on days 1, 8, and 15, and 1 hour infusion of CDDP was administered at a dose of 25 mg/m2 weekly diluted in 500 mL of normal saline to ensure adequate hydration 1 hour before the administration of gemcitabine. Gemcitabine 300mg/m2 will be given by 30-minute intravenous infusion weekly during RT and CRT will be started within 3 weeks after completion of 2 cycles of induction chemotherapy.
  Radiotherapy
  - Total dose of PGTV and PCTV were 55 Gy, 22 fractions and 44 Gy, 22 fractions, respectively.
  Interventions: Radiation: Induction chemotherapy followed by CCRT

INTERVENTIONS:
Radiation: Induction chemotherapy followed by CCRT — Chemotherapy In one cycle (4-weeks), gemcitabine 1,000 mg/m2 will be given by 30-minute intravenous infusion on days 1, 8, and 15, and 1 hour infusion of CDDP was administered at a dose of 25 mg/m2 weekly diluted in 500 mL of normal saline to ensure adequate hydration 1 hour before the administration of gemcitabine. Gemcitabine 300mg/m2 will be given by 30-minute intravenous infusion weekly during CCRT will be started within 3 weeks after completion of 2 cycles of induction chemotherapy
  Radiotherapy
  - Total dose of PGTV and PCTV were 55 Gy, 22 fractions and 44 Gy, 22 fractions, respectively.

SUMMARY:
This phase II trial chose the induction chemotherapy with gemcitabine and cisplatin followed by Chemoradiotherapy (CRT) with gemcitabine to optimize the treatment for pancreas cancer patients with locally advanced disease and the purpose of this trial is to evaluate the efficacy of induction CT with gemcitabine and cisplatin followed by CRT for unresectable pancreatic carcinoma.

DETAILED DESCRIPTION:
The primary endpoint is feasibility and compliance of induction chemotherapy with gemcitabine and cisplatin followed by CRT for locally advanced unresectable pancreatic cancer. Previous studies showed that approximately 20% of patients with locally advanced disease developed the early distant metastasis.[6, 7] Thus, it will be expected that at least 80% of total patients will be eligible for induction chemotherapy after completion of induction chemotherapy. An experimental arm that result a compliance of 80% would merit further study. If the true compliance rate of the patients who will eligible for CRT is ≤ 60%, null hypothesis will be rejected with a power of 80% and a type I error of 5%. Thus, the required number of evaluable patients is 24. Considering the 10% follow-up loss and 20% distant metastasis rate after induction chemotherapy, a total of 34 eligible patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas
* Unresectable locally advanced disease base on institutional standard criteria of unresectability disease following radical surgery. There is no evidence of metastatic disease in the major viscera and no peritoneal seeding
* Patients with biliary or gastroduodenal obstruction must have drainage prior to starting chemoradiation
* All malignant disease must be encompassable within a single irradiation field (15x15cm maximum)
* All patients must have radiographically assessable disease
* No previous irradiation to the planned field
* Age of ≥ 18 years
* performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) score
* Required Entry Laboratory Parameters WBC count ≥ 1,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 100,000/mm3; total bilirubin ≤ 3.0 mg/dL (Patients with elevated bilirubin due to obstruction should be stented and their bilirubin should be decrease ≤ 3.0 mg/dL prior to study entry); creatinine ≤ 3.0 mg/dL
* Oral intake (including J-tube feeding) of ≥ 1,500 calories/day should be maintained.
* Signed informed consent form prior to study entry

Exclusion Criteria:

* There is evidence of metastasis in the major viscera or peritoneal seeding.
* Age of < 18 years
* Previous history of RT adjacent to planned field
* Poor performance status of 2 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* Pregnant or breast feeding status
* Previous history of uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-09-05 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
feasibility and compliance | Up to 1 year
  to evaluate acute and late toxicity of induction chemotherapy with gemcitabine and cisplatin followed by chemoradiotherapy for unresectable pancreatic cancer.

SECONDARY OUTCOMES:
overall survival | Up to 3years until study closed
  To evaluate the impact of induction chemotherapy with gemcitabine and cisplatin followed by concurrent chemoradiotherapy
disease-free survival. | participants will be followed for the duration of disease free, an expected average of 9 months
  To investigate the association between tumor response of induction chemotherapy with gemcitabine and cisplatin followed by concurrent chemoradiotherapy and clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Woo Jin Lee, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No